CLINICAL TRIAL: NCT02486718
Title: A Phase III, Open-Label, Randomized Study to Investigate the Efficacy and Safety of Atezolizumab (Anti-PD-L1 Antibody) Compared With Best Supportive Care Following Adjuvant Cisplatin-Based Chemotherapy in Patients With Completely Resected Stage IB-IIIA Non-Small Cell Lung Cancer
Brief Title: Study to Assess Safety and Efficacy of Atezolizumab (MPDL3280A) Compared to Best Supportive Care Following Chemotherapy in Patients With Lung Cancer [IMpower010]
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO29527; 2014-003205-15 (EudraCT Number); 2023-505981-26-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2015-06-04; First posted 2015-07-01 (Estimated); Results first posted 2025-03-30 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab; Cisplatin; Vinorelbine; Docetaxel; Gemcitabine; Pemetrexed

ARMS (2):
- Atezolizumab (Experimental): Enrollment Phase: Participants will receive four 21-day cycles of cisplatin-based chemotherapy (cisplatin plus either vinorelbine or docetaxel or gemcitabine or pemetrexed [non-squamous cell NSCLC only]), unless unacceptable toxicity, disease relapse, or participant's decision to discontinue occur. Randomization Phase: Participants will receive atezolizumab 1200 milligrams (mg) intravenously (IV) every 3 weeks (Q3W) for sixteen 21-day cycles and will undergo periodic chest X-ray and CT scan.
  Interventions: Drug: Atezolizumab; Drug: Cisplatin; Drug: Vinorelbine; Drug: Docetaxel; Drug: Gemcitabine; Drug: Pemetrexed
- Best Supportive Care (Active Comparator): Enrollment Phase: Participants will receive four 21-day cycles of cisplatin-based chemotherapy (cisplatin plus either vinorelbine or docetaxel or gemcitabine or pemetrexed [non-squamous cell NSCLC only]), unless unacceptable toxicity, disease relapse, or participant's decision to discontinue occur. Randomization Phase: After enrollment phase participants will receive only the best supportive care and will undergo periodic chest X-ray and CT scan.
  Interventions: Drug: Cisplatin; Drug: Vinorelbine; Drug: Docetaxel; Drug: Gemcitabine; Drug: Pemetrexed

INTERVENTIONS:
Drug: Atezolizumab — Participants will receive atezolizumab (1200 mg IV) Q3W for 16 cycles (cycle length=21 days).
  Other Names: MPDL3280A; TECENTRIQ
  Arms: Atezolizumab
Drug: Cisplatin — Participants will receive cisplatin 75 milligrams per square meter (mg/m^2) IV on Day 1 of up to four 21-day cycles.
Drug: Vinorelbine — Participants will receive vinorelbine 30 mg/m^2 IV on Days 1 and 8 of each of the four 21-day cycles.
Drug: Docetaxel — Participants will receive docetaxel 75 mg/m^2 IV on Day 1 of each of the four 21-day cycles.
Drug: Gemcitabine — Participants will receive gemcitabine 1250 mg/m^2 IV on Days 1 and 8 of each of the four 21-day cycles.
Drug: Pemetrexed — Participants will receive pemetrexed 500 mg/m^2 IV on Day 1 of each of the four 21-day cycles. Pemetrexed will be administered only in participants with non-squamous cell NSCLC.

SUMMARY:
This is a Phase III, global, multicenter, open-label, randomized study to compare the efficacy and safety of 16 cycles (1 cycle duration=21 days) of atezolizumab (MPDL3280A) treatment compared with best supportive care (BSC) in participants with Stage IB-Stage IIIA non-small cell lung cancer (NSCLC) following resection and adjuvant chemotherapy, as measured by disease-free survival (DFS) as assessed by the investigator and overall survival (OS). Participants, after completing up to 4 cycles of adjuvant cisplatin-based chemotherapy, will be randomized in a 1:1 ratio to receive atezolizumab for 16 cycles or BSC.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Enrollment Phase

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Histological or cytological diagnosis of Stage IB (tumors greater than or equal to [>/=] 4 centimeters [cm])-IIIA (T2-3 N0, T1-3 N1, T1-3 N2, T4 N0-1) NSCLC (per the Union Internationale Contre le Cancer staging system (UICC)/American Joint Committee on Cancer staging system (AJCC) staging system, 7th edition; Detterbeck et al. 2009)
* Participants must have had complete resection of NSCLC 4-12 weeks (>/=28 days and less than or equal to [</=] 84 days) prior to enrollment and must be adequately recovered from surgery
* If mediastinoscopy was not performed preoperatively, it is required that, at a minimum, mediastinal lymph node systematic sampling will have occurred. Systematic sampling is defined as removal of at least one representative lymph node at specified levels. MLND entails resection of all lymph nodes at those same levels. For a right thoracotomy, sampling or MLND is required at levels 4 and 7 and for a left thoracotomy, levels 5 and/or 6 and 7. Exceptions will be granted if there is clear documentation in the operative report or in a separately submitted addendum by the surgeon of exploration of the required lymph node areas, the participant will be considered eligible if no lymph nodes are found in those areas; if participants have documented N2 disease in one level (per the UICC/AJCC staging system, 7th edition; Detterbeck et al. 2009), not all levels need to be sampled; if the preoperative staging imaging results (contrast computed tomography [CT] and positron emission tomography [PET] scans) do not suggest evidence of disease in the mediastinum, the participant will be considered eligible if N2 nodal sampling is not performed per surgeon's decision
* Eligible to receive a cisplatin-based chemotherapy regimen
* Adequate hematologic and end-organ function
* Women who are not postmenopausal (>/=12 months of non-therapy-induced amenorrhea) or surgically sterile must have a negative serum pregnancy test result within 14 days prior to initiation of cisplatin-based chemotherapy

Inclusion Criteria for Randomized Phase - Women who are not postmenopausal (>/=12 months of non-therapy-induced amenorrhea) or surgically sterile must have a negative serum pregnancy test result within 14 days prior to initiation of atezolizumab or BSC

Exclusion Criteria:

Exclusion Criteria for Enrollment Phase

* Illness or condition that may interfere with a participant's capacity to understand, follow, and/or comply with study procedures
* Pregnant and lactating women
* Treatment with prior systemic chemotherapy: Chemotherapy for early stage of malignancy with curative intent, provided that the last dose received was more than 5 years prior to enrollment and low-dose chemotherapy for non-malignant conditions may be allowed upon approval by the Medical Monitor
* Hormonal cancer therapy or radiation therapy as prior cancer treatment within 5 years before enrollment
* Treatment with any other investigational agent with therapeutic intent within 28 days prior to enrollment
* Participants with hearing impairment
* Known sensitivity to any component of the chemotherapy regimen the participant will be assigned to, or to mannitol
* Prior treatment with cluster of differentiation (CD) 137 (CD137) agonists or immune checkpoint blockade therapies, anti-programmed death-1 (PD-1), and anti programmed death ligand 1 (PD-L1) therapeutic antibodies
* Malignancies other than NSCLC within 5 years prior to randomization, with the exception of those with a negligible risk of metastasis or death (e.g., expected 5-year OS greater than [>] 90 percent [%]) treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated surgically with curative intent, ductal carcinoma in situ treated surgically with curative intent)
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the atezolizumab formulation
* History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis
* Positive test for human immunodeficiency virus (HIV)
* Participants with active hepatitis B (chronic or acute; defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) or hepatitis C
* Active tuberculosis
* Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction, or cerebrovascular accident within the previous 3 months, unstable arrhythmias, or unstable angina
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan
* Prior allogeneic bone marrow transplantation or solid organ transplant
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the participant at high risk from treatment complications
* Known tumor PD-L1 expression status as determined by an immunohistochemistry (IHC) assay from other clinical studies (e.g., participants whose PD-L1 expression status was determined during screening for entry into a study with anti-PD-1 or anti-PD-L1 antibodies but were not eligible are excluded)

Specific Exclusions for Pemetrexed Treatment

- Participants with squamous cell histology

Exclusion Criteria for Randomized Phase

* Signs or symptoms of infection within 14 days prior to randomization (severe infection within 28 days prior to randomization), including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
* Received therapeutic oral or intravenous (IV) antibiotics within 14 days prior to randomization
* Major surgical procedure within 28 days prior to randomization or anticipation of need for a major surgical procedure during the course of the study
* Administration of a live, attenuated vaccine within 4 weeks prior to initiation of study treatment or anticipation that such a live attenuated vaccine will be required during the study
* Treatment with systemic immunostimulatory agents (including but not limited to interferons or interleukin-2) within 4 weeks or 5 half-lives of the drug, whichever is longer, prior to randomization: Prior treatment with cancer vaccines is allowed
* Treatment with systemic corticosteroids or other immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 14 days prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1280 (Actual)
Dates: Start 2015-10-31 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2027-08-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (153):
- United States (32):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - California Cancer Associates for Research & Excellence, Inc., Encinitas, California
  - Compassionate Cancer Care Medical Group, Inc, Fountain Valley, California
  - University of California Los Angeles, Los Angeles, California
  - Kaiser Permanente, Vallejo, California
  - Kaiser Permanente - Walnut Creek, Walnut Creek, California
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Lynn Cancer Institute - West, Boca Raton, Florida
  - University of Miami School of Medicine - Sylvester at Deerfield, Deerfield Beach, Florida
  - SCRI Florida Cancer Specialists North, St. Petersburg, Florida
  - Lewis Hall Singletary Oncology Center, Thomasville, Georgia
  - University of Illinois at Chicago, Chicago, Illinois
  - Illinois Cancer Care, Peoria, Illinois
  - Norton Cancer Institute, Louisville, Kentucky
  - St. Luke's Cancer Institute, Kansas City, Missouri
  - Hematology Oncology Associates of Northern New Jersey, Florham Park, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Valley Hospital, Paramus, New Jersey
  - Overlook Medical Center, Summit, New Jersey
  - Clinical Research Alliance, Lake Success, New York
  - Weill Cornell Medical College, New York, New York
  - Presbyterian Hospital, Charlotte, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care - SCRI, Cincinnati, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University Oncology Associates, Chattanooga, Tennessee
  - Houston Methodist Cancer Center, Houston, Texas
  - Wellmont Medical Associates, Bristol, Virginia
  - Hematology Oncology Associates of Fredericksburg, Inc., Fredericksburg, Virginia
  - MultiCare Regional Cancer Center - Auburn, Auburn, Washington
  - Providence Everett Med Ctr, Everett, Washington
  - Swedish Medical Center, Seattle, Washington
- Australia (2):
  - Townsville Hospital, Douglas, Queensland
  - Cabrini Hospital Malvern, Malvern, Victoria
- Belgium (2):
  - Cliniques Universitaires St-Luc, Brussels
  - CHU de Liège (Sart Tilman), Liège
- China (9):
  - Cancer Institute and Hospital Chinese Academy of Medical Sciences, Beijing
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Anhui Province Cancer Hospital, Hefei
  - Shanghai Chest Hospital, Shanghai
  - Shanghai Pulmonary Hospital, Shanghai
  - Liaoning Provincial Cancer Hospital, Shengyang
  - First Hospital of China Medical University, Shenyang
  - First Affiliated Hospital of Soochow University, Suzhou
- France (7):
  - Centre Hospitalier de Mont de Marsan - Hopital Layne, Mont-de-Marsan
  - Clinique Clémentville, Montpellier
  - Centre Regional de Lutte contre le Cancer Val d Aurelle - Paul Lamarque, Montpellier
  - Centre René Gauducheau Centre de Lutte Contre Le Cancer Nantes Atlantique, Nantes
  - Centre Hospitalier Regional Sud Reunion, Saint-Pierre
  - Centre Hospitalier de Saint-Quentin, Saint-Quentin
  - Hopital d Instruction des Armees de Sainte Anne, Toulon
- Germany (15):
  - Ev.Krankenhaus Bielefeld gGmbH, Bielefeld, North Rhine-Westphalia
  - Evang. Lungenklinik Berlin Klinik für Pneumologie, Berlin
  - Stadtisches Klinikum Braunschweig, Braunschweig
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Krankenhaus Nordwest, Frankfurt am Main
  - LungenClinic Grosshansdorf GmbH, Großhansdorf
  - Lungenklinik Hemer, Hemer
  - Universität Des Saarlandes, Homburg
  - Fachklinik für Lungenerkrankungen, Immenhausen
  - Vincentius-Diakonissen-Kliniken gAG, Karlsruhe
  - Katholisches Klinikum Marienhof, Koblenz Am Rhein
  - Klinikum Bogenhausen, München
  - Gemeinschaftspraxis für Hämatologie und Onkologie, Münster
  - Pius-Hospital Oldenburg, Oldenburg
  - Krankenhaus Barmherzige Bruder Regensburg, Regensburg
- Prince of Wales Hosp, Shatin, Hong Kong
- Hungary (2):
  - University of Pecs, I st Dept of Internal Medicine, Pécs
  - Jasz-Nagykun-Szolnok Megyei Hetenyi Geza Korhaz-Rend.Int., Szolnok
- Israel (5):
  - Rambam Medical Center, Haifa
  - Edith Wolfson Medical Center, Holon
  - Meir Medical Center, Kfar Saba
  - Tel Aviv Sourasky Medical Ctr, Tel Aviv
  - Chaim Sheba Medical Center, Tel Litwinsky
- Italy (12):
  - Ospedale Clinicizzato SS Annunziata, Chieti, Abruzzo
  - Azienda per l'Assistenza Sanitaria N° 5 - Friuli Occidentale, Pordenone, Friuli Venezia Giulia
  - Policlinico Universitario Campus Biomedico Di Roma, Rome, Lazio
  - Asst Papa Giovanni XXIII, Bergamo, Lombardy
  - ASST Spedali Civili di Brescia, Brescia, Lombardy
  - Azienda Sanitaria Ospedaliera S Luigi Gonzaga, Orbassano, Piedmont
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Turin, Piedmont
  - Azienda Ospedaliera Di Rilievo Nazionale E Di Alta Specializzazione Garibaldi, Catania, Sicily
  - Ospedale Santa Chiara, Trento, Trentino-Alto Adige
  - Azienda Ospedaliero Universitaria Pisana, Pisa, Tuscany
  - Ospedale Silvestrini, Perugia, Umbria
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona, Veneto
- Japan (19):
  - Aichi Cancer Center Hospital, Aichi
  - Hyogo Cancer Center, Akashi
  - Juntendo University Hospital, Bunkyō City
  - Tokyo Metropolitan Cancer and Infectious diseases Center Komagome Hospital, Bunkyō City
  - National Cancer Center Hospital, Chūō
  - Kyushu University Hospital, Fukuoka
  - Hiroshima University Hospital, Hiroshima
  - Saitama Cancer Center, Kitaadachi-gun
  - Hospital of the University of Occupational and Environmental Health,Japan, Kitakyushu-shi
  - Kumamoto University Hospital, Kumamoto
  - Kyoto University Hospital, Kyoto
  - Shikoku Cancer Center, Matsuyama
  - Kyorin University Hospital, Mitaka-shi
  - Niigata Cancer Center Hospital, Niigata
  - Okayama University Hospital, Okayama
  - National Hospital Organization Hokkaido Cancer Center, Sapporo
  - Toranomon Hospital, Tokyo
  - Tokyo Medical University Hospital, Tokyo
  - Kanagawa Cancer Center, Yokohama-shi, Asahi-ku
- Netherlands (2):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch, North Brabant
  - St. Antonius Ziekenhuis Nieuwegein, Nieuwegein
- Poland (2):
  - Mazowieckie Centrum Leczenia Chorob Pluc i Gruzlicy, Otwock
  - Wielkopolskie Centrum Pulmonologii i Torakochirurgii w Poznaniu, Poznan
- Portugal (3):
  - Centro Hospitalar E Universitário de Coimbra EPE, Coimbra
  - Instituto Portugues de Oncologia Do Porto Francisco Gentil Epe, Porto
  - Hospital de Sao Joao, Porto
- Oncology Center Sf. Nectarie, Craiova, Romania
- Russia (7):
  - Principal Military Clinical Hospital n.a. N.N. Burdenko, Moscow, Moscow Oblast
  - Leningrad Regional Clinical Hospital, Saint Petersburg, Sankt-Peterburg
  - GBUZ Saint Petersburg Clinical Research Center of Specialized Types of Care (Oncology), Saint Petersburg, Sankt-Peterburg
  - Scientific Research Institute of Oncology n.a. N.N. Petrov, Saint Petersburg, Sankt-Peterburg
  - City Clinical Hospital #1, Novosibirsk
  - Volgograd Regional Clinical Oncology Dispensary, Volgograd
  - Regional Clinical Oncology Hospital, Yaroslavl
- South Korea (2):
  - Chonnam National University Hwasun Hospital, Jeonnam
  - The Catholic University of Korea St. Vincent's Hospital, Suwon
- Spain (14):
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Consorcio Hospitalario Provincial de Castellon, Castellon, Castellon
  - Hospital Universitario Virgen de La Arrixaca, El Palmar, Murcia
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Tenerife
  - Hospital del Mar, Barcelona
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Vall d'Hebron Institute of Oncology (VHIO), Barcelona, Barcelona
  - C.H. Regional Reina Sofia, Córdoba
  - Complejo Hospitalario de Jaen, Jaén
  - Hospital Lucus Augusti, Lugo
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario HM Sanchinarro-CIOCC, Madrid
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
  - Hosp Clinico Univ Lozano Blesa, Zaragoza
- Taiwan (5):
  - Changhua Christian Hospital, Changhua
  - Chang Gung Memorial Hospital Chiayi, Putzui City
  - Taichung Veterans General Hospital, Taichung
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation Linkou Branch, Taoyuan
- Ukraine (9):
  - MI Dnipropetrovsk City Multifield Clinical Hospital 4 of Dnipropetrovsk Regional Council, Dnipropetrovsk, Katerynoslav Governorate
  - Communal Non profit Enterprise Regional Center of Oncology, Kharkiv, Kharkiv Governorate
  - Municipal Institution Odesa Regional Oncology Dispensary, Odesa, KIEV Governorate
  - Municipal Institution SubCarpathian ClinicalOncological Centre, Ivano-Frankivsk, Poltava Governorate
  - Communal Nonprofit Enterprise Podilsky Regional Center Of Oncology OfTheVinnytsia Regional Council, Vinnytsia, Vinnytsia Oblast
  - CE Kryvyi Rih Oncology Dispensary of Dnipropetrovsk Regional Council, Kryvyi Rih
  - Kyiv City Clinical Oncological Center, Kyiv
  - Regional Municipal Institution Sumy Regional Clinical Oncology Dispensary, Sumy
  - MI Zaporizhzhia Regional Clinical Oncological Dispensary Zaporizhzhia SMU Ch of Oncology, Zaporizhzhya
- United Kingdom (2):
  - Colchester General Hospital, Colchester, Essex
  - St Bartholomew's Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Okada M, Sugawara S, Watanabe Y, Saito H, Chen-Yoshikawa TF, Goto Y, Nishio W, Nakagawa S, Hayashi M, Kenmotsu H. IMpower010: 5-Year Outcomes of Atezolizumab in Japanese Patients With Resected Stage IB-IIIA Non-Small Cell Lung Cancer. Cancer Sci. 2025 Dec 19. doi: 10.1111/cas.70297. Online ahead of print. PMID 41416818
- [Derived] Felip E, Altorki N, Zhou C, Vallieres E, Csoszi T, Vynnychenko IO, Goloborodko O, Rittmeyer A, Reck M, Martinez-Marti A, Kenmotsu H, Chen YM, Chella A, Sugawara S, Fu C, Ballinger M, Deng Y, Srivastava MK, Bennett E, Gitlitz BJ, Wakelee HA; IMpower010 Study Investigators. Five-Year Survival Outcomes With Atezolizumab After Chemotherapy in Resected Stage IB-IIIA Non-Small Cell Lung Cancer (IMpower010): An Open-Label, Randomized, Phase III Trial. J Clin Oncol. 2025 Jul 20;43(21):2343-2349. doi: 10.1200/JCO-24-01681. Epub 2025 May 30. PMID 40446184
- [Derived] Zhou C, Srivastava MK, Xu H, Felip E, Wakelee H, Altorki N, Reck M, Liersch R, Kryzhanivska A, Oizumi S, Tanaka H, Hamm J, McCune SL, Bennett E, Gitlitz B, McNally V, Ballinger M, McCleland M, Zou W, Das Thakur M, Novello S. Comparison of SP263 and 22C3 immunohistochemistry PD-L1 assays for clinical efficacy of adjuvant atezolizumab in non-small cell lung cancer: results from the randomized phase III IMpower010 trial. J Immunother Cancer. 2023 Oct;11(10):e007047. doi: 10.1136/jitc-2023-007047. PMID 37903590
- [Derived] Felip E, Altorki N, Zhou C, Vallieres E, Martinez-Marti A, Rittmeyer A, Chella A, Reck M, Goloborodko O, Huang M, Belleli R, McNally V, Srivastava MK, Bennett E, Gitlitz BJ, Wakelee HA. Overall survival with adjuvant atezolizumab after chemotherapy in resected stage II-IIIA non-small-cell lung cancer (IMpower010): a randomised, multicentre, open-label, phase III trial. Ann Oncol. 2023 Oct;34(10):907-919. doi: 10.1016/j.annonc.2023.07.001. Epub 2023 Jul 17. PMID 37467930
- [Derived] Mohindra NA, Patel JD. Top advances in lung cancer, 2021. Cancer. 2022 Oct 1;128(19):3434-3437. doi: 10.1002/cncr.34406. Epub 2022 Aug 10. PMID 35947027
- [Derived] Felip E, Altorki N, Zhou C, Csoszi T, Vynnychenko I, Goloborodko O, Luft A, Akopov A, Martinez-Marti A, Kenmotsu H, Chen YM, Chella A, Sugawara S, Voong D, Wu F, Yi J, Deng Y, McCleland M, Bennett E, Gitlitz B, Wakelee H; IMpower010 Investigators. Adjuvant atezolizumab after adjuvant chemotherapy in resected stage IB-IIIA non-small-cell lung cancer (IMpower010): a randomised, multicentre, open-label, phase 3 trial. Lancet. 2021 Oct 9;398(10308):1344-1357. doi: 10.1016/S0140-6736(21)02098-5. Epub 2021 Sep 20. PMID 34555333

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1280 participants with resectable Stage IB-IIIA non-small cell lung cancer (NSCLC) were enrolled in this study. Participants took part in the study at 227 investigative sites across 22 countries. The study is still ongoing.
Pre-assignment Details: The study consists of 2 phases, an enrollment phase in which participants received up to 4 cycles of adjuvant cisplatin-based chemotherapy followed by randomized phase in which eligible participants were randomized to receive atezolizumab or best supportive care (BSC) i.e.no treatment.
Groups:
- Enrollment Phase: All participants received up to four 21-day cycles of cisplatin-based chemotherapy (cisplatin plus either vinorelbine or docetaxel or gemcitabine or pemetrexed [non-squamous cell NSCLC only] based on investigator's choice), unless unacceptable toxicity, disease relapse, or participant's decision to discontinue occurred.
- Atezolizumab: Participants who did not experience disease recurrence after chemotherapy in enrollment phase received 1200 milligrams (mg) of atezolizumab intravenously (IV) every 3 weeks (Q3W) for sixteen 21-day cycles in the randomization phase.
- Best Supportive Care (BSC): Participants who did not experience disease recurrence after chemotherapy in enrollment phase received no treatment in the randomization phase BSC arm.
Period: Enrollment Phase
Arm/Group | Enrollment Phase | Atezolizumab | Best Supportive Care (BSC)
Started | 1280 | 0 | 0
Enrolled Safety-evaluable Population (Enrolled Safety-evaluable population included all eligible participants who were enrolled in the enrollment phase and who received at least one dose of chemotherapy (cisplatin, vinorelbine, docetaxel, gemcitabine, or pemetrexed), regardless of whether they are subsequently randomized or not.) | 1269 | 0 | 0
Completed | 1005 | 0 | 0
Not Completed | 275 | 0 | 0
Not completed — Death | 19 | 0 | 0
Not completed — Symptomatic deterioration | 1 | 0 | 0
Not completed — Withdrawal by Subject | 86 | 0 | 0
Not completed — Protocol Violation | 18 | 0 | 0
Not completed — Physician Decision | 18 | 0 | 0
Not completed — Reason not provided | 41 | 0 | 0
Not completed — Disease relapse | 54 | 0 | 0
Not completed — Lost to Follow-up | 4 | 0 | 0
Not completed — Adverse Event | 34 | 0 | 0
Period: Randomized Phase
Arm/Group | Enrollment Phase | Atezolizumab | Best Supportive Care (BSC)
Started | 0 | 507 (NOTE: 507 eligible participants were randomized to receive atezolizumab in the randomization phase.) | 498 (NOTE: 498 eligible participants were randomized to receive BSC in the randomization phase.)
Randomized Safety Population (Randomized safety population included all randomized participants who received at least one dose of the study treatment and all randomized participants who were randomized to the control arm and did not receive any dose of atezolizumab but who had at least one post-baseline safety assessment.) | 0 | 495 | 495
Completed | 0 | 0 | 0
Not Completed | 0 | 507 | 498
Not completed — Withdrawal by Subject | 0 | 44 | 47
Not completed — Protocol Violation | 0 | 2 | 0
Not completed — Physician Decision | 0 | 0 | 3
Not completed — Lost to Follow-up | 0 | 5 | 11
Not completed — Disease Relapse | 0 | 1 | 0
Not completed — Death | 0 | 154 | 155
Not completed — Ongoing | 0 | 301 | 282

BASELINE CHARACTERISTICS:
Population: Enrolled population was defined as all eligible participants who were enrolled in the enrollment phase, regardless if they are subsequently randomized or not.
Arm/Group | Enrollment Phase
Number analyzed (Participants) | 1280
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 427
  Male | 853
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18
  Not Hispanic or Latino | 1219
  Unknown or Not Reported | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 307
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 8
  White | 935
  More than one race | 1
  Unknown or Not Reported | 27

OUTCOME MEASURES:

1. Primary Outcome: Disease-Free Survival (DFS) in Intent-to-treat (ITT) Population
Description: DFS was defined as the time from randomization to the first recurrence of NSCLC or occurrence of new primary NSCLC as determined by the investigator or death, whichever occurs first. Kaplan-Meier methodology was used to estimate the median DFS for each treatment arm.
Time Frame: Up to 95 months
Population: Randomized ITT population was defined as all randomized participants with resected Stage IB [tumors ≥ 4 centimetres (cm)]-IIIA NSCLC whether or not the participant received the assigned treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab | Best Supportive Care (BSC)
Number analyzed (Participants) | 507 | 498
months | 65.6 [52.4 to NA] — The upper limit of the 95% confidence interval (CI) was not estimable due to insufficient number of participants with events. | 47.8 [37.0 to 65.8]
Statistical Analysis 1: Comparison: Atezolizumab vs Best Supportive Care (BSC); Test type: Superiority — Stratified Analysis; p = 0.0683, Log Rank; Hazard Ratio (HR) = 0.848, 95% CI 2-sided [0.710 to 1.013]

2. Primary Outcome: DFS in All Randomized Stage II-IIIA Population
Description: DFS was defined as the time from randomization to the first recurrence of NSCLC or occurrence of new primary NSCLC as determined by the investigator or death, whichever occurs first. DFS was analyzed in participants with disease stage II-IIIA. Kaplan-Meier methodology was used to estimate the median DFS for each treatment arm.
Time Frame: Up to 95 months
Population: Stage II-IIIA population was defined as all randomized participants with extent of disease as either Stage II or Stage IIIA, and is a subset of the ITT population. Randomized ITT population was defined as all randomized participants with resected Stage IB (tumors ≥ 4 cm)-IIIA NSCLC whether or not the participant received the assigned treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab | Best Supportive Care (BSC)
Number analyzed (Participants) | 442 | 440
months | 57.4 [42.2 to NA] — The upper limit of the 95% CI was not estimable due to insufficient number of participants with events. | 40.8 [31.4 to 57.1]
Statistical Analysis 1: Comparison: Atezolizumab vs Best Supportive Care (BSC); Test type: Superiority — Stratified Analysis; Hazard Ratio (HR) = 0.830, 95% CI 2-sided [0.691 to 0.998]

3. Primary Outcome: DFS in the Programmed Death-ligand 1 (PD-L1) SP263 ≥ 1% Tumor Cell (TC) Subpopulation Within the Stage II-IIIA Population
Description: DFS was defined as the time from randomization to the first recurrence of NSCLC or occurrence of new primary NSCLC as determined by the investigator or death, whichever occurs first. DFS was analyzed in PD-L1 ≥1% subpopulation within the Stage II-IIIA population. Kaplan-Meier methodology was used to estimate the median DFS for each treatment arm.
Time Frame: Up to 95 months
Population: PD-L1 subpopulation, defined as ≥1% TC expression by the SP263 immunohistochemistry (IHC) assay, included Stage II-IIIA population with valid PD-L1 SP263 measurement at baseline. Stage II-IIIA population included all randomized participants with extent of disease as either Stage II or Stage III, & is a subset of ITT population. Randomized ITT population included all randomized participants with resected Stage IB (tumors ≥ 4 cm)-IIIA NSCLC whether the participant received the assigned treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab | Best Supportive Care (BSC)
Number analyzed (Participants) | 248 | 228
months | 68.5 [51.8 to NA] — The upper limit of the 95% CI was not estimable due to insufficient number of participants with events. | 37.3 [30.1 to 57.8]
Statistical Analysis 1: Comparison: Atezolizumab vs Best Supportive Care (BSC); Test type: Superiority — Stratified Analysis; Hazard Ratio (HR) = 0.704, 95% CI 2-sided [0.545 to 0.910]

4. Secondary Outcome: Overall Survival (OS) in the ITT Population
Description: OS was defined as the time from randomization to death from any cause.
Time Frame: Baseline up to death from any cause (up to approximately 126 months)
Reporting Status: Not Posted, anticipated posting 2028-08

5. Secondary Outcome: Disease-free Rate at Year 3 in ITT Population
Description: DFS rate was defined as percentage of participants who were disease-free at Year 3. The DFS rate was estimated by the Kaplan-Meier methodology for each treatment arm. Percentages have been rounded off to the nearest decimal.
Time Frame: Year 3
Population: Randomized ITT population was defined as all randomized participants with resected Stage IB (tumors ≥ 4 cm)-IIIA NSCLC whether or not the participant received the assigned treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab | Best Supportive Care (BSC)
Number analyzed (Participants) | 507 | 498
percentage of participants | 61.43 [57.09 to 65.77] | 55.45 [50.95 to 59.95]
Statistical Analysis 1: Comparison: Atezolizumab vs Best Supportive Care (BSC); Test type: Superiority; Difference in event-free rates = 5.98, 95% CI 2-sided [-0.28 to 12.23]

6. Secondary Outcome: Disease-free Rate at Year 3 in All Randomized Stage II-IIIA Population
Description: DFS rate was defined as percentage of participants who were disease-free at Year 3. DFS rate was analyzed in participants with disease stage II-IIIA. The DFS rate was estimated by the Kaplan-Meier methodology for each treatment arm. Percentages have been rounded off to the nearest decimal.
Time Frame: Year 3
Population: Stage II-IIIA population was defined as all randomized participants with extent of disease as either Stage II or Stage III, and is a subset of the ITT population. Randomized ITT population was defined as all randomized participants with resected Stage IB (tumors ≥ 4 cm)-IIIA NSCLC whether or not the participant received the assigned treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab | Best Supportive Care (BSC)
Number analyzed (Participants) | 442 | 440
percentage of participants | 59.30 [54.61 to 63.98] | 52.64 [47.83 to 57.46]
Statistical Analysis 1: Comparison: Atezolizumab vs Best Supportive Care (BSC); Test type: Superiority; Difference in event-free rates = 6.65, 95% CI 2-sided [-0.06 to 13.36]

7. Secondary Outcome: Disease-free Rate at Year 3 in PD-L1 (SP263 ≥ 1% TC) Subpopulation Within the Stage II-IIIA Population
Description: DFS rate was defined as percentage of participants who were disease-free at Year 3. DFS rate was analyzed in PD-L1 subpopulation within the Stage II-IIIA population. The DFS rate was estimated by the Kaplan-Meier methodology for each treatment arm. Percentages have been rounded off to the nearest decimal.
Time Frame: Year 3
Population: PD-L1 subpopulation, defined as ≥ 1% TC expression by the SP263 IHC assay, included Stage II-IIIA population with valid PD-L1 SP263 measurement at baseline. Stage II-IIIA population included all randomized participants with extent of disease as either Stage II or Stage III, & is a subset of ITT population. Randomized ITT population included all randomized participants with resected Stage IB (tumors ≥ 4 cm)-IIIA NSCLC whether the participant received the assigned treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab | Best Supportive Care (BSC)
Number analyzed (Participants) | 248 | 228
percentage of participants | 62.72 [56.54 to 68.90] | 52.05 [45.35 to 58.75]
Statistical Analysis 1: Comparison: Atezolizumab vs Best Supportive Care (BSC); Test type: Superiority; Difference in event-free rates = 10.67, 95% CI 2-sided [1.56 to 19.79]

8. Secondary Outcome: Disease-free Rate at Year 5 in ITT Population
Description: DFS rate was defined as percentage of participants who were disease-free at Year 5. The DFS rate was estimated by the Kaplan-Meier methodology for each treatment arm. Percentages have been rounded off to the nearest decimal.
Time Frame: Year 5
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab | Best Supportive Care (BSC)
Number analyzed (Participants) | 507 | 498
percentage of participants | 51.96 [47.45 to 56.46] | 46.48 [41.91 to 51.05]
Statistical Analysis 1: Comparison: Atezolizumab vs Best Supportive Care (BSC); Test type: Superiority; Difference in event-free rates = 5.48, 95% CI 2-sided [-0.94 to 11.90]

9. Secondary Outcome: Disease-free Rate at Year 5 in All Randomized Stage II-IIIA Population
Description: DFS rate was defined as percentage of participants who were disease-free at Year 5. DFS rate was analyzed in participants with disease stage II-IIIA. The DFS rate was estimated by the Kaplan-Meier methodology for each treatment arm. Percentages have been rounded off to the nearest decimal.
Time Frame: Year 5
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab | Best Supportive Care (BSC)
Number analyzed (Participants) | 442 | 440
percentage of participants | 49.28 [44.47 to 54.10] | 44.40 [39.57 to 49.24]
Statistical Analysis 1: Comparison: Atezolizumab vs Best Supportive Care (BSC); Test type: Superiority; Difference in event-free rates = 4.88, 95% CI 2-sided [-1.94 to 11.70]

10. Secondary Outcome: Disease-free Rate at Year 5 in PD-L1 (SP263 ≥ 1% TC) Subpopulation Within the Stage II-IIIA Population
Description: DFS rate was defined as percentage of participants who were disease-free at Year 5. DFS rate was analyzed in PD-L1 subpopulation within the Stage II-IIIA population. The DFS rate was estimated by the Kaplan-Meier methodology for each treatment arm. Percentages have been rounded off to the nearest decimal.
Time Frame: Year 5
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab | Best Supportive Care (BSC)
Number analyzed (Participants) | 248 | 228
percentage of participants | 53.15 [46.69 to 59.61] | 42.69 [36.00 to 49.38]
Statistical Analysis 1: Comparison: Atezolizumab vs Best Supportive Care (BSC); Test type: Superiority; Difference in event-free rates = 10.46, 95% CI 2-sided [1.16 to 19.76]

11. Secondary Outcome: DFS in the PD-L1 (SP263 ≥ 50% TC) Subpopulation Within the Stage II-IIIA Population
Description: DFS was defined as the time from randomization to the first recurrence of NSCLC or occurrence of new primary NSCLC as determined by the investigator or death, whichever occurs first. DFS was analyzed in PD-L1 subpopulation within the Stage II-IIIA population. Kaplan-Meier methodology was used to estimate the median DFS for each treatment arm.
Time Frame: Up to 95 months
Population: PD-L1 subpopulation, defined as ≥50% TC expression by the SP263 IHC assay, included Stage II-IIIA population with valid PD-L1 SP263 measurement at baseline. Stage II-IIIA population included all randomized participants with extent of disease as either Stage II or Stage III, & is a subset of ITT population. Randomized ITT population included all randomized participants with resected Stage IB (tumors ≥ 4 cm)-IIIA NSCLC whether the participant received the assigned treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab | Best Supportive Care (BSC)
Number analyzed (Participants) | 115 | 114
months | NA [NA to NA] — The median and the 95% CI was not estimable due to insufficient number of participants with events. | 41.1 [29.7 to NA] — The upper limit of the 95% CI was not estimable due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Atezolizumab vs Best Supportive Care (BSC); Test type: Superiority — Stratified Analysis; Hazard Ratio (HR) = 0.503, 95% CI 2-sided [0.332 to 0.761]

12. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a participant when administered a pharmaceutical product regardless of the causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom/disease temporally associated with the use of an investigational product, whether or not considered related to the investigational product.
Time Frame: Up to 12 years
Reporting Status: Not Posted, anticipated posting 2028-08

13. Secondary Outcome: Percentage of Participants With Anti-Therapeutic Antibodies (ATAs) to Atezolizumab
Description: The percentage of ATA (Also called anti-drug antibodies (ADA))-positive participants after drug administration were determined for participants exposed to atezolizumab. For determining post-baseline incidence, participants were considered to be ADA-positive if they were ADA-negative or had missing data at baseline but developed an ADA response following study drug exposure, or if they were ADA-positive at baseline and the titer of 1 or more post-baseline samples was at least 0.60 titer units (t.u.) greater than the baseline titer result.
Time Frame: Predose (Hour 0) on Day 1 of Cycles 2, 3, 4, 8, 16 (Cycle length = 21 days), at treatment discontinuation (TD) (up to 12 months), 120 days after last atezolizumab administration (up to 16 months)
Population: ADA evaluable population was defined as all randomized participants who received at least one dose of atezolizumab and who have at least one post-baseline ADA result.
Measure: Number; unit: percentage of participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 487
percentage of participants | 31.2

14. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Atezolizumab
Time Frame: 30 min post-infusion on Day 1 of Cycle 1 (Cycle length = 21 days)
Population: PK-evaluable population was defined as all randomized participants who received any dose of the study treatment and who have evaluable pharmacokinetic samples. Overall number analyzed is the number of participants with data available for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/millilitres (μg/ml)
Arm/Group | Atezolizumab
Number analyzed (Participants) | 451
micrograms/millilitres (μg/ml) | 367 (124)

15. Secondary Outcome: Minimum Serum Concentration (Cmin) at Steady-State Within a Dosing Interval of Atezolizumab
Time Frame: Prior to infusion on Day 1 of Cycles 1, 2, 3, 4, 8, 16 (Cycle length = 21 days), at study discontinuation visit (up to 12 months), Day 120 post last dose of atezolizumab (up to 16 months)
Population: PK-evaluable population was defined as all randomized participants who received any dose of the study treatment and who have evaluable pharmacokinetic samples. Number analyzed is the number of participants with data available for analyses at the specified timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/ml
Arm/Group | Atezolizumab
Number analyzed (Participants) | 493
μg/ml
  Cycle 1 Day 1: number analyzed (Participants) | 451
  Cycle 1 Day 1 | 367 (123.5)
  Cycle 2 Day 1: number analyzed (Participants) | 446
  Cycle 2 Day 1 | 87.8 (79.3)
  Cycle 3 Day 1: number analyzed (Participants) | 436
  Cycle 3 Day 1 | 141 (58.4)
  Cycle 4 Day 1: number analyzed (Participants) | 419
  Cycle 4 Day 1 | 170 (57.6)
  Cycle 8 Day 1: number analyzed (Participants) | 353
  Cycle 8 Day 1 | 222 (40.6)
  Cycle 16 Day 1: number analyzed (Participants) | 300
  Cycle 16 Day 1 | 221 (87.3)
  Treatment Discontinuation Visit: number analyzed (Participants) | 404
  Treatment Discontinuation Visit | 148 (221.8)
  Day 120 Post Last Dose of Atezolizumab: number analyzed (Participants) | 352
  Day 120 Post Last Dose of Atezolizumab | 8.58 (794.8)

ADVERSE EVENTS:
Time Frame: Up to 95 months
Description: Enrolled safety-evaluable population included patients in enrollment phase & received at least 1 dose of chemo. Randomized safety-evaluable population included randomized patients who received at least 1 dose of atezo & randomized patients who were randomized to control arm & did not receive any dose of atezo but had at least 1 post-baseline safety assessment, regardless of their assigned treatment at randomization. All-cause mortality reported for deaths that occurred during study based on ITT.
Arm/Group | Enrollment Phase | Best Supportive Care (BSC) | Atezolizumab
All-Cause Mortality (participants affected / at risk) | 19/1269 | 155/495 | 154/495
Serious Adverse Events (participants affected / at risk) | 259/1269 | 42/495 | 88/495
Other Adverse Events (participants affected / at risk) | 1153/1269 | 227/495 | 358/495
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrollment Phase (N=1269) | Best Supportive Care (BSC) (N=495) | Atezolizumab (N=495)
Anaemia (Blood and lymphatic system disorders) | 8 (8) | 0 (0) | 1 (1)
Sarcoidosis of lymph node (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0) | 2 (2)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Hypopituitarism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Secondary adrenocortical insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Death (General disorders) | 3 (3) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 3 (3) | 1 (1) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 6 (6)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (2)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Contrast media reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 2 (2) | 0 (0) | 1 (1)
Immune-mediated adverse reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Sarcoidosis (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (2)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Encephalitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Otitis media chronic (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pleural infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 18 (18) | 5 (5) | 8 (9)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 5 (5) | 0 (0) | 2 (2)
Septic shock (Infections and infestations) | 2 (2) | 1 (1) | 2 (2)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0) | 2 (2)
Viral myocarditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Comminuted fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Prescribed overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Urethral stricture traumatic (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 2 (2) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Intestinal metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Langerhans' cell histiocytosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of head and neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Urinary tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Axonal neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Demyelinating polyneuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Encephalitis autoimmune (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Intracranial haematoma (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 5 (5) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 2 (3) | 0 (0)
Dissociative disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Hallucination, visual (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 6 (6) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Adnexal torsion (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (3)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (5)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 22 (22) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 2 (2) | 0 (0)
Thrombophlebitis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Agranulocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Bone marrow failure (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 38 (42) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Myelosuppression (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 13 (14) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Otolithiasis (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 12 (12) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Varices oesophageal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 10 (12) | 0 (0) | 0 (0)
Asthenia (General disorders) | 2 (2) | 0 (0) | 0 (0)
Device related thrombosis (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0)
Malaise (General disorders) | 4 (6) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Performance status decreased (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bacterial abdominal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bacterial diarrhoea (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Device related sepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Intervertebral discitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Stitch abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vascular device infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (4) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (4) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 9 (10) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 4 (4) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Autonomic neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Hypotonia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Intercostal neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Device occlusion (Product Issues) | 1 (1) | 0 (0) | 0 (0)
Catatonia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0)
Bronchial fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 4 (4) | 0 (0) | 0 (0)
Granulomatosis with polyangiitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Subclavian vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrollment Phase (N=1269) | Best Supportive Care (BSC) (N=495) | Atezolizumab (N=495)
Anaemia (Blood and lymphatic system disorders) | 357 (422) | 30 (30) | 37 (47)
Hyperthyroidism (Endocrine disorders) | 7 (7) | 3 (3) | 33 (36)
Hypothyroidism (Endocrine disorders) | 3 (3) | 3 (3) | 54 (61)
Diarrhoea (Gastrointestinal disorders) | 181 (226) | 9 (12) | 36 (54)
Nausea (Gastrointestinal disorders) | 660 (1032) | 16 (16) | 31 (44)
Asthenia (General disorders) | 234 (301) | 14 (15) | 37 (45)
Fatigue (General disorders) | 269 (309) | 11 (14) | 33 (41)
Pyrexia (General disorders) | 75 (86) | 11 (14) | 60 (67)
Nasopharyngitis (Infections and infestations) | 25 (26) | 50 (65) | 33 (44)
Upper respiratory tract infection (Infections and infestations) | 27 (33) | 12 (14) | 37 (43)
Alanine aminotransferase increased (Investigations) | 52 (57) | 16 (17) | 54 (71)
Aspartate aminotransferase increased (Investigations) | 43 (47) | 16 (16) | 54 (67)
Blood creatinine increased (Investigations) | 85 (113) | 15 (15) | 29 (36)
Arthralgia (Musculoskeletal and connective tissue disorders) | 36 (41) | 26 (35) | 52 (65)
Headache (Nervous system disorders) | 77 (90) | 20 (22) | 28 (39)
Cough (Respiratory, thoracic and mediastinal disorders) | 93 (101) | 46 (55) | 66 (84)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 64 (64) | 32 (33) | 31 (35)
Pruritus (Skin and subcutaneous tissue disorders) | 22 (26) | 3 (3) | 51 (55)
Rash (Skin and subcutaneous tissue disorders) | 54 (58) | 5 (7) | 48 (58)
Leukopenia (Blood and lymphatic system disorders) | 84 (128) | 5 (6) | 5 (10)
Neutropenia (Blood and lymphatic system disorders) | 338 (568) | 5 (5) | 21 (33)
Thrombocytopenia (Blood and lymphatic system disorders) | 67 (94) | 6 (9) | 9 (11)
Tinnitus (Ear and labyrinth disorders) | 69 (75) | 6 (6) | 6 (8)
Constipation (Gastrointestinal disorders) | 317 (389) | 9 (10) | 24 (27)
Vomiting (Gastrointestinal disorders) | 248 (361) | 9 (9) | 20 (27)
Malaise (General disorders) | 66 (94) | 2 (2) | 5 (5)
Neutrophil count decreased (Investigations) | 187 (367) | 3 (3) | 9 (10)
Platelet count decreased (Investigations) | 73 (108) | 1 (1) | 10 (12)
White blood cell count decreased (Investigations) | 111 (221) | 1 (1) | 6 (7)
Decreased appetite (Metabolism and nutrition disorders) | 305 (421) | 7 (7) | 23 (28)
Dizziness (Nervous system disorders) | 70 (74) | 15 (15) | 18 (20)
Dysgeusia (Nervous system disorders) | 95 (106) | 1 (1) | 2 (2)
Insomnia (Psychiatric disorders) | 75 (80) | 6 (6) | 21 (21)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 89 (142) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 181 (183) | 10 (10) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsorâ€™s intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2024-05-24): https://cdn.clinicaltrials.gov/large-docs/18/NCT02486718/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-30): https://cdn.clinicaltrials.gov/large-docs/18/NCT02486718/SAP_001.pdf